CLINICAL TRIAL: NCT00303329
Title: Extension Study of Iron Chelation Therapy With Deferasirox in β-thalassemia and Other Patients With Rare Chronic Anemia and Transfusional Iron Overload
Brief Title: Extension Study of Iron Chelation Therapy With Deferasirox in β-thalassemia and Rare Chronic Anemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0108E1
Record Dates: First submitted 2005-10-14; First posted 2006-03-16 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Anemia; Hemosiderosis
Keywords: β-thalassemia; rare chronic anemia; iron overload; deferasirox; chronic anemias; transfusional hemosiderosis
MeSH Terms: conditions — Anemia; Hemosiderosis; Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deferasirox (Experimental): Deferasirox daily oral dose between 5-40 mg/kg/day
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Deferasirox available as 125 mg, 250 mg or 500 mg tablets
  Other Names: ICL670

SUMMARY:
A 1-year randomized Phase II core trial was conducted to investigate the efficacy of deferasirox in regularly transfused patients with β-thalassemia and other rare chronic anemia 2 years of age and older. Patients who successfully completed the main trial may continue in the extension trial to receive chelation therapy with deferasirox for up to 3 years. Extension was prolonged to 4 years.

The objective of this study is to assess the long-term safety and efficacy of deferasirox in these patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients completed the planned 12-month core study
* Female patients who have reached menarche and who are sexually active must use double-barrier contraception, oral contraceptive plus barrier contraceptive, or must have undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation
* Written informed consent obtained from the patient and/or legal guardian on the patient's behalf in accordance with the national legislation

Exclusion Criteria:

* Pregnant or breast feeding patients

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2004-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (5):
  - Children's Hospital and Research center at Oakland, Oakland, California
  - Stanford Hospital, Stanford, California
  - Childres's Hospital Boston, Boston, Massachusetts
  - New York Presbyterian Hospital, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Belgium (5):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Toronto
- France (4):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Troyes
- Germany (3):
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Ulm
- Italy (8):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Brindisi
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Rome
  - Novartis Investigative Site, Torino
- Novartis Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- β-thalassemia Patients; Rare Anemias Patients: Deferasirox (5-40 mg/kg/day)
Period: Overall Study
Arm/Group | β-thalassemia Patients | Rare Anemias Patients
Started | 85 | 99
Completed | 50 | 37
Not Completed | 35 | 62
Not completed — Adverse Event | 7 | 14
Not completed — Abnormal Laboratory Values | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 9 | 2
Not completed — Condition no longer requires study drug | 0 | 8
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 9 | 15
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative problems | 1 | 0
Not completed — Death | 2 | 12
Not completed — Stopped at end of core | 3 | 9
Not completed — Stopped at end of extension 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | β-thalassemia Patients | Rare Anemias Patients | Total
Number analyzed (Participants) | 85 | 99 | 184
Age Continuous [Mean (Standard Deviation); unit: years] | 24.7 (10.03) | 43.7 (26.13) | 35.0 (22.4)
Age, Customized [Number; unit: participants]
  <6 years | 2 | 9 | 11
  Between 6 and 11 years | 5 | 6 | 11
  Between 12 and 15 years | 8 | 5 | 13
  Between 16 and 49 years | 69 | 30 | 99
  Between 50 and 64 years | 1 | 19 | 20
  >=65 years | 0 | 30 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 91
  Male | 42 | 51 | 93
Region of Enrollment [Number; unit: participants]
  United States | 15 | 21 | 36
  France | 9 | 11 | 20
  Canada | 12 | 6 | 18
  Belgium | 4 | 12 | 16
  Germany | 2 | 23 | 25
  United Kingdom | 12 | 0 | 12
  Italy | 31 | 26 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) or Deaths
Description: Safety was assessed using reports of adverse events of all participants in this study. Serious adverse events are those events that resulted in death, were life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: Core study Baseline to the end of the study (up to 60 months)
Population: The safety analysis set comprised all participants who received at least one dose of deferasirox during either the core or extension studies.
Measure: Number; unit: Participants
Arm/Group | β-thalassemia Patients | Rare Anemias Patients
Number analyzed (Participants) | 85 | 99
Participants
  Adverse Events | 85 | 99
  Serious Adverse Events | 36 | 50
  Deaths | 2 | 12

2. Secondary Outcome: The Change in Liver Iron Content (LIC) as Assessed by Liver Biopsy at Baseline to the End of the Study
Description: Liver iron concentration was monitored at the start of the core study, the end of the core study, and then at the end of the extension study. High-risk participants, like participants with rare anemia, were excluded from any further potential liver biopsy, except if required and justified by the Investigator for the general care of the participant.
Time Frame: Core study Baseline to end of extension study (up to 60 months)
Population: The full analysis Set (FAS) comprised all participants who received at least one dose of deferasirox during either the core or extension studies.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | β-thalassemia Patients | Rare Anemias Patients
Number analyzed (Participants) | 55 | 42
mg Fe/g dw | -5.17 (11.659) | -5.10 (7.756)

3. Secondary Outcome: The Absolute Change in Liver Iron Content (LIC) as Assessed by Superconducting Quantum Interference Device (SQUID) From Baseline to End of Study
Description: Liver iron concentration was monitored at the end of the core study and then at the end of the extension study. High-risk participants, like participants with rare anemia, were excluded from any further potential liver biopsy, except if required and justified by the Investigator for the general care of the participant. Pediatric participants or participants with a medical contraindication to liver biopsy were allowed the use of SQUID in the extension study.
Time Frame: Core study Baseline to end of extension study (up to 60 months)
Population: The FAS comprised all participants who received at least one dose of deferasirox during either the core or extension studies.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | β-thalassemia Patients | Rare Anemias Patients
Number analyzed (Participants) | 15 | 33
mg Fe/g dw | 0.19 (8.577) | -2.04 (4.521)

4. Secondary Outcome: The Absolute Change in Serum Ferritin (μg/L) Levels From Baseline to the End of the Study
Description: Serum ferritin was monitored monthly and the dose of deferasirox was increased or decreased in steps of 5 to 10 mg/kg/day up to a maximum of 40 mg/kg/day if appropriate, every 3 months. If serum ferritin fell to 500 ng/mL or lower on two consecutive study visits, an interruption of treatment until serum ferritin was more than 500 ng/mL was considered.
Time Frame: Core study Baseline to end of extension study (up to 60 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | β-thalassemia Patients | Rare Anemias Patients
Number analyzed (Participants) | 85 | 96
μg/L
  Baseline | 4320.6 (2881.08) | 3268.8 (2082.60)
  End of Study | 3708.2 (3018.10) | 2896.0 (2597.22)
  Absolute Change | -612.4 (2520.87) | -382.2 (2325.41)

ADVERSE EVENTS:
Groups:
- Beta-thalassemia; Rare Anemias: Deferasirox (5-40 mg/kg/day)
Arm/Group | Beta-thalassemia | Rare Anemias
Serious Adverse Events (participants affected / at risk) | 36/85 | 50/99
Other Adverse Events (participants affected / at risk) | 84/85 | 96/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Beta-thalassemia (N=85) | Rare Anemias (N=99)
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Primary hypogonadism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Catheter related complication (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Chills (General disorders) | 0 | 2
Drug withdrawal syndrome (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 12
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 2
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis yersinia (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 0 | 2
Meningitis viral (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 5
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 5
Septic shock (Infections and infestations) | 0 | 3
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Coma (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 3
Illusion (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Testicular disorder (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Beta-thalassemia (N=85) | Rare Anemias (N=99)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 1
Palpitations (Cardiac disorders) | 12 | 8
Tachycardia (Cardiac disorders) | 12 | 6
Ear pain (Ear and labyrinth disorders) | 10 | 6
Tinnitus (Ear and labyrinth disorders) | 6 | 0
Vertigo (Ear and labyrinth disorders) | 6 | 6
Vision blurred (Eye disorders) | 5 | 1
Abdominal discomfort (Gastrointestinal disorders) | 7 | 3
Abdominal distension (Gastrointestinal disorders) | 10 | 5
Abdominal pain (Gastrointestinal disorders) | 32 | 31
Abdominal pain upper (Gastrointestinal disorders) | 30 | 13
Constipation (Gastrointestinal disorders) | 23 | 14
Diarrhoea (Gastrointestinal disorders) | 40 | 50
Dyspepsia (Gastrointestinal disorders) | 9 | 7
Gastritis (Gastrointestinal disorders) | 1 | 7
Gingival bleeding (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 36 | 34
Toothache (Gastrointestinal disorders) | 12 | 3
Vomiting (Gastrointestinal disorders) | 23 | 36
Asthenia (General disorders) | 14 | 19
Chest pain (General disorders) | 19 | 9
Fatigue (General disorders) | 17 | 18
Influenza like illness (General disorders) | 9 | 4
Malaise (General disorders) | 5 | 4
Oedema (General disorders) | 2 | 8
Oedema peripheral (General disorders) | 7 | 12
Pyrexia (General disorders) | 39 | 36
Hepatomegaly (Hepatobiliary disorders) | 4 | 5
Seasonal allergy (Immune system disorders) | 8 | 6
Bronchitis (Infections and infestations) | 9 | 20
Ear infection (Infections and infestations) | 7 | 3
Gastroenteritis (Infections and infestations) | 14 | 17
Influenza (Infections and infestations) | 14 | 15
Nasopharyngitis (Infections and infestations) | 33 | 26
Oral herpes (Infections and infestations) | 3 | 8
Otitis media (Infections and infestations) | 3 | 6
Pharyngitis (Infections and infestations) | 26 | 4
Rhinitis (Infections and infestations) | 21 | 12
Sinusitis (Infections and infestations) | 3 | 6
Tonsillitis (Infections and infestations) | 9 | 8
Tooth abscess (Infections and infestations) | 7 | 1
Tooth infection (Infections and infestations) | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 23 | 16
Urinary tract infection (Infections and infestations) | 10 | 10
Viral infection (Infections and infestations) | 5 | 2
Viral upper respiratory tract infection (Infections and infestations) | 10 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 3
Procedural pain (Injury, poisoning and procedural complications) | 14 | 3
Transfusion reaction (Injury, poisoning and procedural complications) | 13 | 13
Blood creatinine increased (Investigations) | 16 | 19 — This is the number patients with clinically notable increases in serum creatinine, not just patients with increases.
Cardiac murmur (Investigations) | 5 | 5
Transaminases increased (Investigations) | 3 | 5
Weight decreased (Investigations) | 2 | 5
Anorexia (Metabolism and nutrition disorders) | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 9
Dizziness (Nervous system disorders) | 5 | 8
Headache (Nervous system disorders) | 45 | 34
Paraesthesia (Nervous system disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 6 | 4
Depression (Psychiatric disorders) | 11 | 8
Insomnia (Psychiatric disorders) | 8 | 7
Dysuria (Renal and urinary disorders) | 7 | 3
Proteinuria (Renal and urinary disorders) | 5 | 3
Renal failure (Renal and urinary disorders) | 0 | 6
Dysmenorrhoea (Reproductive system and breast disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Erythema (Skin and subcutaneous tissue disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 9
Rash (Skin and subcutaneous tissue disorders) | 14 | 13
Rash pruritic (Skin and subcutaneous tissue disorders) | 7 | 1
Haematoma (Vascular disorders) | 1 | 5
Hypertension (Vascular disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.